CLINICAL TRIAL: NCT02819687
Title: A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single- and Multiple-Ascending Doses of RDX5791 in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RDX5791 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RDX5791-101
Record Dates: First submitted 2016-06-07; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Phase I; Healthy; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- RDX5791 10mg QD (SAD phase) (Experimental): 10mg of RDX5791 administered once daily PO fasting
  Interventions: Drug: RDX5791; Drug: Placebo
- RDX5791 50mg QD (SAD phase) (Experimental): 50mg of RDX5791 administered once daily PO fasting
  Interventions: Drug: RDX5791; Drug: Placebo
- RDX5791 150mg QD (SAD phase) (Experimental): 150mg of RDX5791 administered once daily PO fasting
  Interventions: Drug: RDX5791; Drug: Placebo
- RDX5791 450mg QD (SAD phase) (Experimental): 450mg of RDX5791 administered once daily PO fasting
  Interventions: Drug: RDX5791; Drug: Placebo
- RDX5791 900mg QD (SAD phase) (Experimental): 900mg of RDX5791 administered once daily PO fasting
  Interventions: Drug: RDX5791; Drug: Placebo
- RDX5791 3mg QD (MAD phase) (Experimental): 3mg of RDX5791 administered once daily PO fasting
  Interventions: Drug: RDX5791; Drug: Placebo
- RDX5791 10mg QD (MAD phase) (Experimental): 10mg of RDX5791 administered once daily PO fasting
  Interventions: Drug: RDX5791; Drug: Placebo
- RDX5791 30 mg QD (MAD phase) (Experimental): 30mg of RDX5791 administered once daily PO fasting
  Interventions: Drug: RDX5791; Drug: Placebo
- RDX5791 100 mg QD (MAD phase) (Experimental): 100mg of RDX5791 administered once daily PO fasting
  Interventions: Drug: RDX5791; Drug: Placebo

INTERVENTIONS:
Drug: RDX5791
  Other Names: Tenapanor; AZD1722
Drug: Placebo

SUMMARY:
A Phase I, single-center, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single-and multiple-ascending doses of RDX5791 in healthy male and female subjects.

DETAILED DESCRIPTION:
In the single-ascending dose (SAD), 5 separate cohorts received RDX5791 at various doses once po fasting. Each cohort of 8 subjects (6 RDX5791, 2 placebo) received a diet standardized fro Na+ content wile in the clinical pharmacology unit (CPU).

The PK data from the 50-mg dose and the safety data from the 150-mg dose of the SAD study were evaluated prior to proceeding with the multiple-ascending dose (MAD) phase. Doses of RDX5791 are 3, 10, 30, and 100 mg administered once daily po fasting. Four cohorts of 10 subjects each (8 RDX5791, 2 placebo) received a diet standardized for Na+ content while in the CPU.

Safety assessments including clinical assessment and vital signs, clinical laboratory evaluations, ECGs, and AE monitoring were performed at regular intervals. Plasma was collected at regular intervals for PK analysis. The PD assessment included stool frequency and consistency, as well as changes in urinary Na+ excretion. All bowel movements were collected and analyzed for Na+ content outside this study protocol.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 29.9 kg/m², inclusive
* Females must be of non-childbearing potential; If of child-bearing potential, must have negative pregnancy test and confirm the use of one of the appropriate means of contraception
* Males must agree to use appropriate methods of barrier contraception or have documented surgical sterilization

Exclusion Criteria:

* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the GI tract
* Any surgery on the small intestine or colon, excluding appendectomy
* Loose stools (Bristol Stool Form Score of 6 or 7) ≥2 days in the past 7 days
* Hepatic dysfunction ([ALT] or [AST]) >1.5 times the upper limit of normal or renal impairment
* Any evidence of or treatment of malignancy, excluding non-melanomatous malignancies of the skin
* Use of diuretic medications, medications that are known to affect stool consistency and/or GI motility
* Use of an investigational agent within 30 days prior to Day -2
* Positive virology, alcohol, or drugs of abuse test during screening
* Use of any prescription medication within 7 days before admission to the CPU
* Have had significant blood loss (>450 mL) or have donated 1 or more units of blood or plasma within 8 weeks prior to study entry

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | 7 days
  serum chemistry and hematology, ECGs, and clinical signs and symptoms

SECONDARY OUTCOMES:
Pharmacokinetics of RDX5791 | 7 days
  blood levels of drug
Urinary and fecal sodium levels | 7 days
  to assess the pharmacodynamics of RDX5791
Urinary and fecal phosphorus levels | 7 days
  to assess the pharmacodynamics of RDX5791

CONTACTS AND LOCATIONS:
Overall Officials: David P. Rosenbaum, Ph.D, Study Chair — Ardelyx, Inc.

REFERENCES:
- [Derived] Rosenbaum DP, Yan A, Jacobs JW. Pharmacodynamics, Safety, and Tolerability of the NHE3 Inhibitor Tenapanor: Two Trials in Healthy Volunteers. Clin Drug Investig. 2018 Apr;38(4):341-351. doi: 10.1007/s40261-017-0614-0. PMID 29363027